CLINICAL TRIAL: NCT01087476
Title: Phase 2 Double-blind, Randomized, Placebo Controlled Clinical Trial for the Prevention of Oral Mucositis Using Sub-microbial Doses of Doxycycline Hyclate in Patients With Acute Leukemia Receiving Induction Chemotherapy
Brief Title: Double-blind-randomized,Placebo Controlled Trial for Chemotherapy-associated Oral Mucositis Using Doxycycline Hyclate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Metropolitan Autonomous University (Other)
Collaborators: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Dr. Velia A. Ramírez-Amador, Universidad Autonoma Metropolitana-Xochimilco
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: MetropolitanAU
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Mucositis
Keywords: oral mucositis; chemotherapy; acute leukemia; salivary flow.
MeSH Terms: conditions — Mucositis; Stomatitis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- doxycycline hyclate (Experimental): Patients will be randomly assigned to receive either a sub-microbial dose of doxycycline hyclate or placebo (50 mg per day), immediately before the initiation of induction chemotherapy and daily during the following 21 days after chemotherapy.
  Interventions: Drug: Doxycycline hyclate

INTERVENTIONS:
Drug: Doxycycline hyclate — Sub-microbial dose of Doxycycline hyclate or placebo (50 mg per day), immediately before the initiation of induction chemotherapy and daily during the following 21 days after chemotherapy.
  Other Names: Doryx; Doxine; Vibramycin

SUMMARY:
Background. Mucositis is a complication of chemotherapy with no effective treatment. Aim.To evaluate the efficacy of sub-microbial doses of doxycycline hyclate in preventing the development of oral mucositis in patients with acute leukemia (AL) treated with induction chemotherapy.

Hypothesis. Doxycycline hyclate administration in sub-microbial dosage will reduce the incidence of oral mucositis in patients with AL who receive induction chemotherapy.

Methods. Double-blind, randomized, placebo-controlled clinical trial. At the Cancer National Institute (INCan), adult patients (> 18 years of age) with acute leukemia of recent diagnosis, scheduled to receive induction chemotherapy will be enrolled in the study. Written informed consent from the patients will be obtained preceding inclusion in the study.

At baseline and 3-times per week, during 21-days, patients will have an oral examination performed using the Oral Mucositis Assessment Scale (OMAS), oral pain, difficulty to swallow, and salivary flow measurements will be recorded.

A sample size of 164 subjects has been calculated, 74 subjects in each arm of the study. The primary end point of this study to evaluate the efficacy will be the proportion of patients treated with doxycycline or placebo without oral lesions associated with OM, during the 21 days of follow-up. Efficacy will be evaluated if the proportion of complete response (CR) is significantly higher than the proportion of events in the placebo group. Additional secondary endpoints will be the partial resolution of the oral lesions, the incidence of infections and the mortality in the study groups during the 21 days of follow-up. Results will be analyzed by using Chi-squared test and Wilcoxon-Mann-Whitney rank sum test.

DETAILED DESCRIPTION:
Background. Mucositis is a complication of chemotherapy with no effective treatment.

Aim.To evaluate the efficacy of sub-microbial doses of doxycycline hyclate in preventing the development of oral mucositis in patients with acute leukemia (AL) treated with induction chemotherapy.

Hypothesis. Doxycycline hyclate administration in sub-microbial dosage will reduce the incidence of oral mucositis in patients with AL who receive induction chemotherapy.

Methods. Double-blind, randomized, placebo-controlled clinical trial. At the Cancer National Institute (INCan), adult patients (> 18 years of age) with acute leukemia of recent diagnosis, scheduled to receive induction chemotherapy will be enrolled in the study. Written informed consent from the patients will be obtained preceding inclusion in the study.

Stratification according to the type of acute leukemia (myeloblastic and lymphoblastic) will be done. Random number tables will be used with balance for every four subjects; coded boxes will be utilized to preserve double blinding. Patients will be randomly assigned to receive either a sub-microbial dose of doxycycline hyclate or placebo (50 mg per day), immediately before the initiation of induction chemotherapy and daily during the following 21 days after chemotherapy.

At baseline and 3-times per week, during 21-days, patients will have an oral examination performed using the Oral Mucositis Assessment Scale (OMAS). Also oral pain and difficulty to swallow will be recorded using a visual analogue scale. Also in each visit, salivary flow measurements (Schirmer's test modified version) will be done.

The OMAS system is a validated index that evaluates the severity of oral mucositis by measuring the degree of ulceration/pseudomembrane and erythema in nine sites of the oral mucosa (upper and lower lip, right and left inner cheek, right and left ventral and lateral tongue, floor of the mouth, soft palate/fauces and hard palate). At each site, erythema is evaluated using a 3-point scale (0=none, 1=mild/moderate, 2=severe), and ulceration/pseudomembrane formation is evaluated using a 4-point scale (0=none, 1=cumulative surface area <1 cm2, 2=cumulative surface area 1-3 cm2, 3=cumulative surface area >3 cm2). The value of OMAS will be obtained by summing the erythema and ulceration/pseudomembrane sub-scores at each site and then averaging these scores across the affected sites.

In order to rule out oral candidosis (OC), definitive diagnosis of OC requires the identification of pseudohyphae in exfoliative cytology samples stained with periodic acid Schiff. Likewise, the clinical diagnosis of herpes simplex virus (HSV) induced oral lesions will be confirmed by the virus-infected cells demonstrated in cytologic smears stained with Papanicolaou, and/or a clinical response to systemic antiviral therapy with acyclovir.

A sample size of 164 subjects has been calculated, 74 subjects in each arm of the study. This estimate is based in the incidence of OM that is higher than 40% in patients with AL, and considering its reduction to half (20%), assuming an alpha value of 0.05 (one-sided) and a minimum statistical power of 0.80.

The efficacy primary end point of this study will be the proportion of patients treated with doxycycline or placebo without oral lesions associated with OM, in the 21 days of follow-up. Efficacy will be evaluated if the proportion of complete response (CR) is significantly higher than the proportion of events in the placebo group. Additional secondary endpoints will be the partial resolution of the oral lesions, the incidence of infections and the mortality in the study groups during the 21 days of follow-up.

Statistical analysis. Results will be analysed by using Chi-squared test and Wilcoxon-Mann-Whitney rank sum test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years of age) with acute leukemia of recent diagnosis,scheduled to receive induction chemotherapy.
* Capacity to give written informed consent.
* Ability to attend the follow-up visits.

Exclusion Criteria:

* Patients with allergy or intolerance to tetracyclines
* Patients with acute or chronic renal insufficiency (basal blood creatinine >1.9 mg/dl)
* Patients with the contraindication for the oral administration of drugs.
* Patients with active septic processes or considered resolved in less than 7 days before the start of chemotherapy.
* Patients who required tetracycline administration in the 28 days previous to randomization.
* Adult patients with acute leukemia schedule to undergo stem-cell transplantation in the following two weeks.
* Adult patients with hematological cancer with previous radiotherapy that may affect the salivary glands.
* Inability to authorize a written informed consent.

Exclusion criteria

* Patients who start chemotherapy before 12 hours of the assigned treatment.
* Patients who have received less than 10 doses (5 days) of the assigned treatment.
* Requirement to receive ergot derivates.
* Patients who require the administration of acitretin/isotretinoin/tretinoin
* Patients that receive photosensitive drugs during the study period (hydroxyquinone/retinoids or methoxsalen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Complete response | At baseline and 3-times per week, during 21-days after chemotherapy.
  Complete response will be evaluated through the OMAS score.

SECONDARY OUTCOMES:
Partial resolution of oral lesions, incidence of infections and mortality. | At baseline and 3-times per week, during 21-days after chemotherapy.
  Partial response will be evaluated through the OMAS score. The incidence of infections and the mortality in the study groups during the 21 days of follow-up.To confirm the diagnosis of oral candidosis (OC), the identification of pseudohyphae in exfoliative cytology samples stained with periodic acid Schiff, will be necessary. The clinical diagnosis of herpes simplex virus (HSV) induced will be confirmed by the virus-infected cells demonstrated in cytologic smears stained with Papanicolaou, and/or a clinical response to systemic antiviral therapy with acyclovir.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Ponce de Leon, MD, Study Director — Instituto Nacional de Ciencias Médicas y Nutrición
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Ramirez-Amador V, Anaya-Saavedra G, Crespo-Solis E, Camacho EI, Gonzalez-Ramirez I, Ponce-de-Leon S. Prospective evaluation of oral mucositis in acute leukemia patients receiving chemotherapy. Support Care Cancer. 2010 May;18(5):639-46. doi: 10.1007/s00520-009-0708-1. Epub 2009 Aug 6. PMID 19655176